CLINICAL TRIAL: NCT02433444
Title: Computer Aided, Non-invasive, Acoustic Gastrointestinal Surveillance (AGIS) in Post-ERCP Pancreatitis (PEP)
Brief Title: Computer Aided, Non-invasive, Acoustic Gastrointestinal Surveillance in Post-ERCP Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Elham Afghani, Assistant Director,Clinical Pancreatology, Cedars-Sinai Medical Center
Other Study IDs: Pro00039663
Record Dates: First submitted 2015-04-23; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatitis
Keywords: Biosensing Techniques
MeSH Terms: conditions — Pancreatitis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving ERCP: Patients receiving Endoscopic retrograde cholangiopancreatography (ERCP) at Cedars-Sinai Medical Center.
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — ERCP's performed at Cedars-Sinai Medical Center.

SUMMARY:
In this study, the investigators aim to distinguish patients with Post-Endoscopic retrograde cholangiopancreatography (ERCP) Pancreatitis (PEP) vs. those without PEP based on difference in pre- vs. post-ERCP measurements of AGIS-derived intestinal rates (IR). Based on the clinical observation that many patients with PEP develop ileus following ERCP, the investigators hypothesize that patients who develop PEP will exhibit lower IR following ERCP, and therefore a larger difference in pre- vs. post-ERCP IR.

DETAILED DESCRIPTION:
This will be a prospective case series in 100 patients presenting to Cedars Sinai Medical Center who undergo Endoscopic retrograde cholangiopancreatography (ERCP).

The investigators will place the AGIS sensor on each patient enrolled in the study, 30 minutes prior to procedure. The investigators will continuously record AGIS acoustic signals from T-30 minutes to the time that they leave the hospital, either on discharge from the Post-Anesthesia Care Unit or discharge from hospitalization, with the option to discontinue if clinically required or requested by the provider or patient. Acoustic signal will be evaluated, and intestinal motility events will be calculated; however, this data will not be used to make decisions regarding clinical care. Physicians and nurses will not be made aware of the AbStats readings.These measurements are solely observational. Patients will be managed according to standard-of-care practice.

Routinely, patients are kept in the post-operative unit after their procedure, for one hour. Those with pain are examined by a physician and the decision is made to admit for observation to monitor for complications of ERCP, or to discharge home. The patients who are discharged home from procedure will be followed by telephone surveys every day for 2 days post procedure to determine if they have developed symptoms suggestive of PEP. If so, they will be asked to go to the closest urgent care or emergency department for further evaluation. Those who are admitted for observations post procedure will be followed for signs or symptoms of PEP which includes meeting 2 of 3 criteria: Abdominal pain, amylase/lipase >3 times the upper limit of normal 24 hours after procedure, and/or imaging consistent with pancreatitis.

The AGIS multi-sensor wireless abdominal monitoring system includes low profile acoustic sensors that are applied to the anterior abdominal wall with Tegaderm and monitors sounds emanating from the GI tract. The acoustic sensors continuously and non-invasively monitor and capture audio signals representing GI and abdominal wall function. The captured data is recorded in a synchronized manner from two sensors, each placed 3cm on either side of the umbilicus.

After a patient's participation in the study is complete, the investigators will analyze the AbStats readings and the their clinical outcomes to observe if correlations exist between patients with lower intestinal rates and those who develop PEP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patient of Cedars-Sinai Medical Center scheduled for outpatient ERCP to be performed by one of the study investigators/treating physicians
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide consent
* Transfer patients
* Cognitive inability to follow directions to maintain sensors in place
* Unable to place abdominal sensors on patients
* Abdominal cellulitis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will recruit patients presenting to Cedars-Sinai Medical Center for outpatient ERCP to be performed by one of the study investigators/treating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intestinal Rate | Participants will be followed for the duration of their hospital stay, an expected average of 4 days, and for 2 days after hospital discharge.
  Count of motility events (as measured by AGIS) per minute

CONTACTS AND LOCATIONS:
Overall Officials: Elham Afghani, MD, Principal Investigator — Cedars-Sinai Medical Center

REFERENCES:
- [Background] Freeman ML, DiSario JA, Nelson DB, Fennerty MB, Lee JG, Bjorkman DJ, Overby CS, Aas J, Ryan ME, Bochna GS, Shaw MJ, Snady HW, Erickson RV, Moore JP, Roel JP. Risk factors for post-ERCP pancreatitis: a prospective, multicenter study. Gastrointest Endosc. 2001 Oct;54(4):425-34. doi: 10.1067/mge.2001.117550. PMID 11577302
- [Background] Rieger H, Runkel N, Sproder J, Buhr HJ. [Different mechanisms in intestinal paralysis in edematous and necrotizing pancreatitis of the rat]. Langenbecks Arch Chir Suppl Kongressbd. 1998;115(Suppl I):409-12. German. PMID 14518287
- [Background] Augustyniak P. Wearable wireless heart rate monitor for continuous long-term variability studies. J Electrocardiol. 2011 Mar-Apr;44(2):195-200. doi: 10.1016/j.jelectrocard.2010.11.014. PMID 21353066
- [Background] Shambroom JR, Fabregas SE, Johnstone J. Validation of an automated wireless system to monitor sleep in healthy adults. J Sleep Res. 2012 Apr;21(2):221-30. doi: 10.1111/j.1365-2869.2011.00944.x. Epub 2011 Aug 22. PMID 21859438
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837